CLINICAL TRIAL: NCT06343922
Title: Effects Of Oral Motor Facilitation Technique And Traditional Exercises On Drooling And Feeding Skills Of Children With Cerebral Palsy
Brief Title: Oral Motor Facilitation Technique And Traditional Exercises on Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sadaf Riphah
Record Dates: First submitted 2023-12-26; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy (CP)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Group 1 will receive exercises by using oral motor facilitation technique protocol three times a week Group 2 will receive traditional oral motor exercises three times per week
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral motor facilitation technique group (Experimental): Exercise by using OMFT protocol will be given in the order of warming up technique, key point technique and application technique for 30 min a day.
  Interventions: Behavioral: oral motor facilitation technique group
- traditional oral motor exercises group (Other): Traditional exercises of lips, cheeks, tongue and jaws will be provided for 30 min a day and 3 days/week
  Interventions: Other: traditional oral motor exercises group

INTERVENTIONS:
Behavioral: oral motor facilitation technique group — oral motor facilitation technique
  Arms: oral motor facilitation technique group
Other: traditional oral motor exercises group — traditional oral motor exercises
  Arms: traditional oral motor exercises group

SUMMARY:
Cerebral palsy is a motor disorder caused by the damage to the developing brain. Feeding and swallowing difficulties are common in children with cerebral palsy (CP). Poor postural control and oral motor dysfunction results in extended feeding time, frequent coughing, choking and excessive drooling affecting their health and quality of life. The brain damage in CP is permanent that cannot be fixed however different oral motor exercises, oral facial facilitation and oral sensorimotor interventions are widely used for drool reduction and feeding difficulties in children with CP. Spastic cerebral palsy is one of most prevalent type of CP that is characterized by increased tone and stiffness of muscles. This research will be conducted to evaluate the comparative effects of oral motor facilitation technique (OMFT) and traditional oral motor exercises on drooling and feeding skills of children with spastic CP. OMFT is a complete protocol with a combination of techniques to deal with oral motor difficulties This study will be a randomized control trial. A total number of 12 children with Spastic cerebral palsy ( GMFS III-V) both male/female, between age range 3-12 and with feeding difficulties will be included in the study. Children with cerebral palsy and other co morbidities, seizures, risk of aspiration and who are on tube feeding will be excluded. Participants will be randomly allocated to two groups, either Group A (receiving OMFT) or Group B (receiving traditional oral motor exercise). Baseline scores will be recorded by using standardized tools OMAS for oral motor skill during feeding and DIS for drool severity with the consent of authors. Therapeutic sessions will be scheduled 3 days per week and 30 min a day for each group. The effects of interventions on drooling and feeding skills will be assessed after 8 and 16 weeks of sessions. Recorded data of all variables will be analyzed by using statistical package for social sciences (SPSS) for Windows Software, version 21.

DETAILED DESCRIPTION:
Cerebral palsy is a motor disorder caused by the damage to the developing brain. Feeding and swallowing difficulties are common in children with cerebral palsy (CP). Poor postural control and oral motor dysfunction results in extended feeding time, frequent coughing, choking and excessive drooling affecting their health and quality of life. The brain damage in CP is permanent that cannot be fixed however different oral motor exercises, oral facial facilitation and oral sensorimotor interventions are widely used for drool reduction and feeding difficulties in children with CP. Spastic cerebral palsy is one of most prevalent type of CP that is characterized by increased tone and stiffness of muscles. This research will be conducted to evaluate the comparative effects of oral motor facilitation technique (OMFT) and traditional oral motor exercises on drooling and feeding skills of children with spastic CP. OMFT is a complete protocol with a combination of techniques to deal with oral motor difficulties This study will be a randomized control trial. A total number of 12 children with Spastic cerebral palsy ( GMFS III-V) both male/female, between age range 3-12 and with feeding difficulties will be included in the study. Children with cerebral palsy and other co morbidities, seizures, risk of aspiration and who are on tube feeding will be excluded. Participants will be randomly allocated to two groups, either Group A (receiving OMFT) or Group B (receiving traditional oral motor exercise). Baseline scores will be recorded by using standardized tools OMAS for oral motor skill during feeding and DIS for drool severity with the consent of authors. Therapeutic sessions will be scheduled 3 days per week and 30 min a day for each group. The effects of interventions on drooling and feeding skills will be assessed after 8 and 16 weeks of sessions. Recorded data of all variables will be analyzed by using statistical package for social sciences (SPSS) for Windows Software, version 21.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy
* Type: spastic CP
* Severity level :GMFCS (gross motor function classification scale) level III to V, with head and neck control problems
* With feeding and oral motor difficulties
* Gender male/female
* Age: 3-10 years
* No past history of receiving OMFT

Exclusion Criteria:

* CP children with other co morbidities or syndromes
* risk of aspiration
* children on tube feeding or with seizures
* children with craniofacial anomalies

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Change in Drooling | 16 weeks
  Change in drooling of CP children will be measured by using "Drooling Impact scale", a quantitative tool to evaluate the effects of intervention on drool control. It is a 10 item scale with 10 point scoring level from 0 (no impact at all) to 10 (severe impact) to quantify the impact of intervention.
Change in feeding skills | 16 weeks
  A change in oral motor skills during feeding after intervention will be evaluated by using "Oral Motor Assessment Scale", a seven item/variable scale and each variable scores from 0 (not functional ) to 3 ( normal function). At the end total score is measured and an increase in score shows the improvement in feeding skills.

CONTACTS AND LOCATIONS:
Overall Officials: Nazia Mumtaz, PhD, Principal Investigator — Riphah International University
Locations (1):
- Mobilty Quest, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Widman-Valencia ME, Gongora-Meza LF, Rubio-Zapata H, Zapata-Vazquez RE, Lizama EV, Salomon MR, Estrella-Castillo D. Oral Motor Treatment Efficacy: Feeding and Swallowing Skills in Children with Cerebral Palsy. Behav Neurol. 2021 Oct 25;2021:6299462. doi: 10.1155/2021/6299462. eCollection 2021. PMID 34733374
- [Background] Min KC, Seo SM, Woo HS. Effect of oral motor facilitation technique on oral motor and feeding skills in children with cerebral palsy : a case study. BMC Pediatr. 2022 Nov 3;22(1):626. doi: 10.1186/s12887-022-03674-8. PMID 36324103
- [Background] Abd-Elmonem AM, Saad-Eldien SS, Abd El-Nabie WA. Effect of oral sensorimotor stimulation on oropharyngeal dysphagia in children with spastic cerebral palsy: a randomized controlled trial. Eur J Phys Rehabil Med. 2021 Dec;57(6):912-922. doi: 10.23736/S1973-9087.21.06802-7. Epub 2021 May 7. PMID 33960181
- [Background] Reid SM, Johnson HM, Reddihough DS. The Drooling Impact Scale: a measure of the impact of drooling in children with developmental disabilities. Dev Med Child Neurol. 2010 Feb;52(2):e23-8. doi: 10.1111/j.1469-8749.2009.03519.x. Epub 2009 Oct 15. PMID 19843155
- [Background] Ortega Ade O, Ciamponi AL, Mendes FM, Santos MT. Assessment scale of the oral motor performance of children and adolescents with neurological damages. J Oral Rehabil. 2009 Sep;36(9):653-9. doi: 10.1111/j.1365-2842.2009.01979.x. Epub 2009 Jul 15. PMID 19627455